CLINICAL TRIAL: NCT00812253
Title: Intensive Glycemic Control for Congestive Heart Failure Exacerbation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kathleen Dungan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Kathleen Dungan, Assistant Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007H0197; 1K23DK080891-01A1 (NIH)
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Results first posted 2014-08-07 (Estimated); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Congestive Heart Failure; Diabetes Mellitus
Keywords: Heart failure; Hyperglycemia; Hospital; Diabetes Mellitus
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous Insulin (Experimental)
  Interventions: Drug: Intravenous insulin
- Subcutaneous Insulin (Active Comparator): Basal bolus insulin (4 injections per day)
  Interventions: Drug: Subcutaneous insulin

INTERVENTIONS:
Drug: Intravenous insulin — Half of subjects will receive insulin through the intravenous route while the other half will receive 4 injections per day.
  Arms: Intravenous Insulin
Drug: Subcutaneous insulin — Half of subjects will receive insulin through the intravenous route while the other half will receive 4 injections per day.
  Arms: Subcutaneous Insulin

SUMMARY:
Patients with heart failure often have high blood sugar (glucose).

DETAILED DESCRIPTION:
Patients with heart failure often have high blood sugar. High glucose contributes to severe hospital complications and even death. Studies suggest that heart failure patients who have high glucose or diabetes do not live as long as patients with normal glucose. In this study, we will determine whether normalizing blood sugars using intravenous insulin short-term will improve outcomes in patients hospitalized for congestive heart failure. We enrolled patients with severe heart failure and randomly assigned them into 2 groups. We used intravenous (given through the vein) insulin to lower blood sugar levels in group 1, and insulin injections in group 2. We determined whether intravenous insulin improved hospital length of stay, rates of readmission, inflammatory markers, and cardiovascular tests that predict mortality in patients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* Admitted (less than 48 hours) to the OSU Ross Heart Hospital with worsening heart failure
* Hyperglycemia or diabetes. Hyperglycemia is defined as blood glucose greater than 150 mg/dL on at least 2 occasions separated by at least 4 hours apart, insulin use, or HbA1c >6.5%.

Exclusion Criteria:

* Type 1 diabetes
* Receiving comfort care measures only
* Hospital stay expected to be less than 2 days
* Pregnancy
* Prisoners
* Participation in the study on prior hospitalizations
* Acute myocardial infarction within 3 months
* End stage renal or liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2009-01; Primary Completion 2013-09 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Dungan, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intravenous Insulin (IV): Intravenous insulin: In patients assigned to intravenous (IV) insulin, SQ basal insulin was discontinued and IV insulin was started at 21:00 on the day of enrollment. Patients continued to receive subcutaneous prandial insulin. All patients receiving IV insulin were managed using our hospital's universal nursing run guideline, which has a target glucose of 6.1-8.3 mmol/l. Patients were transitioned from the infusion after 48 hours using approximately 70% of the estimated basal insulin infusion requirement with 4 hours of overlap.
- Subcutaneous Insulin: Basal bolus insulin (4 injections per day) In subjects who were insulin naïve, the total daily dose of insulin was calculated as 0.4 or 0.5 unit/kg if the enrollment glucose was <11.1 mmol/l or >11.1 mmol/l respectively. In subjects who were not insulin naive, the total insulin dose was calculated as 100% or 120% of the total daily insulin dose at admission in subjects with an enrollment glucose of <11.1 mmol/l or >11.1 mmol/l respectively. Basal and prandial insulin were administered in approximately equal total daily doses with correction dosing and adjustments based upon a published algorithm. The target glucose range was 5.6-8.3 mmol/l.
Period: Overall Study
Arm/Group | Intravenous Insulin (IV) | Subcutaneous Insulin
Started | 32 | 42
Completed | 26 | 39
Not Completed | 6 | 3
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline population consists of patients with available study data.
Groups:
- Intravenous (IV) Insulin: Intravenous (IV) insulin: In patients assigned to IV insulin, SQ basal insulin was discontinued and IV insulin was started at 21:00 on the day of enrollment. Patients continued to receive subcutaneous prandial insulin. All patients receiving IV insulin were managed using our hospital's universal nursing run guideline, which has a target glucose of 6.1-8.3 mmol/l. Patients were transitioned from the infusion after 48 hours using approximately 70% of the estimated basal insulin infusion requirement with 4 hours of overlap.
- Subcutaneous (SQ) Insulin: Basal bolus insulin (4 injections per day) In subjects who were insulin naïve, the total daily dose of insulin was calculated as 0.4 or 0.5 unit/kg if the enrollment glucose was <11.1 mmol/l or >11.1 mmol/l respectively. In subjects who were not insulin naive, the total insulin dose was calculated as 100% or 120% of the total daily insulin dose at admission in subjects with an enrollment glucose of <11.1 mmol/l or >11.1 mmol/l respectively. Basal and prandial insulin were administered in approximately equal total daily doses with correction dosing and adjustments based upon a published algorithm. The target glucose range was 5.6-8.3 mmol/l.
- Total: Total of all reporting groups
Arm/Group | Intravenous (IV) Insulin | Subcutaneous (SQ) Insulin | Total
Number analyzed (Participants) | 26 | 39 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (10) | 63 (12) | 62 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 13 | 21
  Male | 18 | 26 | 44
Region of Enrollment [Number; unit: participants]
  United States | 26 | 39 | 65
Preserved ejection fraction [Number; unit: participants] — Preserved ejection fraction was defined as greater than 50%
  participants
    Preserved Ejection Fraction | 6 | 11 | 17
    Reduced Ejection Fraction | 20 | 28 | 48
HbA1c [Mean (Standard Deviation); unit: Percentage of hemoglobin] | 8.4 (2.0) | 7.7 (1.4) | 8.0 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Hospital Length of Stay
Description: Duration of hospitalization in days
Time Frame: Days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Intravenous (IV) Insulin | Subcutaneous (SQ) Insulin
Number analyzed (Participants) | 26 | 39
days | 7 [5 to 11] | 8 [5 to 12]

2. Secondary Outcome: Hospital Readmission
Description: All-cause hospital readmission at 30 days after discharge
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Intravenous (IV) Insulin | Subcutaneous (SQ) Insulin
Number analyzed (Participants) | 26 | 39
participants
  Readmitted | 7 | 15
  Not readmitted | 19 | 24

3. Secondary Outcome: Heart Rate Variability
Description: High frequency (HF) Heart rate variability (HRV). HRV was assessed with a Bionex system (Mindware, Gahanna, OH). The electrocardiogram was performed in the standard lead II configuration and impedance cardiography was performed using a standard tetrapolar arrangement. Measures were performed at baseline and each morning (0800-1000 hour) during and following the intervention for 7 minutes each. Software (Mindware, Gahanna, OH) was used to derive HF HRV. The middle five minutes of the recordings were scored minute by minute and the first suitable1 minute period was used for calculation. Five minute epochs were not feasible due to an unexpectedly high frequency of ectopy. One minute intervals allow calculation of HF (parasympathetic tone) but not low frequency (combination of sympathetic and parasympathetic tone).
Time Frame: 72 hours
Population: Subjects with medical devices, conditions that preclude measurement of HRV such as arrhythmias, or technical problems could not be analyzed.
Measure: Median (Inter-Quartile Range); unit: ms^2
Arm/Group | Intravenous (IV) Insulin | Subcutaneous (SQ) Insulin
Number analyzed (Participants) | 12 | 10
ms^2 | 5.1 [2.26 to 14.8] | 20.7 [4.92 to 312.9]

4. Secondary Outcome: Change in Quality of Life
Description: Change in Quality of Life questionnaire measured from baseline (enrollment) to 30 days following discharge. The questionnaire is a self-administered disease-specific questionnaire for patients with HF, comprising 21 items rated on six-point Likert scales, representing different degrees of impact of HF on health related quality of life, from 0 (none) to 5 (very much). It provides a total score (range 0-105, from best to worst HRQoL),
Time Frame: 30 day
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravenous (IV) Insulin | Subcutaneous (SQ) Insulin
Number analyzed (Participants) | 19 | 35
units on a scale | -22.4 (22.0) | -22.6 (26.3)

5. Secondary Outcome: Brain Natriuretic Peptide (BNP)
Description: Brain natriuretic peptide (BNP) was measured at day 3
Time Frame: 72 hours
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Intravenous (IV) Insulin | Subcutaneous (SQ) Insulin
Number analyzed (Participants) | 26 | 39
pg/ml | 794 [168 to 1090] | 356 [192 to 910]

6. Secondary Outcome: Cardiac Output
Description: Cardiac output measured using impedance cardiography at 72 hours.
Time Frame: 72 hours
Population: Patients without data due to medical devices, conditions that preclude measurement of PEP such as arrhythmias, or technical problems.
Measure: Mean (Standard Deviation); unit: liter/min
Arm/Group | Intravenous (IV) Insulin | Subcutaneous (SQ) Insulin
Number analyzed (Participants) | 13 | 11
liter/min | 10.3 (9.3) | 8.6 (3.5)

ADVERSE EVENTS:
Time Frame: 72 hours after enrollment
Arm/Group | Intravenous (IV) Insulin | Subcutaneous (SQ) Insulin
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/39
Other Adverse Events (participants affected / at risk) | 9/26 | 3/39
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intravenous (IV) Insulin (N=26) | Subcutaneous (SQ) Insulin (N=39)
Hypoglycemia (Endocrine disorders) | 9 | 3 — Hypoglycemia defined as a blood glucose value 3.9<mmol/L

LIMITATIONS AND CAVEATS:
HRV and impedance data were limited due to medical devices, conditions that preclude measurement of HRV such as arrhythmias, or technical problems (N=2). The remainder of missing data were due to early hospital discharge.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No